CLINICAL TRIAL: NCT06547411
Title: Effects of Different Ventilation Modes on Intracranial Pressure and Carbon Dioxide Partial Pressure During Bariatric Surgery: a Prospective, Randomized, Controlled Study
Brief Title: Effects of Different Anesthesia Machine Modalities on Bariatric Surgery Patients: a Prospective Randomized Controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yu-Long Jia (Other)
Collaborators: Inner Mongolia Baogang Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other)
Responsible Party: Sponsor-Investigator, Yu-Long Jia, Principal Investigator, Inner Mongolia University of Science and Technology
Organization: Inner Mongolia University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MER-068
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-08

CONDITIONS: Ventilation; Bariatric Surgery; Intracranial Pressure; Carbon Dioxide
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PC Ventilation mode group (Experimental): Group I patients received mechanical ventilation using the PC mode. The anesthetic machine (MAQUET Flow-I, Italy) parameters were set as follows: The inspiratory pressure (Pins) was adjusted to maintain an end-tidal carbon dioxide concentration (ETCO2) of 4.0-5.0 kPa. Pure oxygen and air were utilized at 0.3 L/min each, with an oxygen content of 41%.
  Interventions: Device: PC Ventilation mode
- VC Ventilation mode group (Experimental): Group II patients received mechanical ventilation in VC mode. The tidal volume during regulated breathing was determined based on the ideal body weight (IBW): 6-8 ml/kg (IBW for males: 50 + 0.91 × (height [cm] - 152.4); IBW for females: 45.5 + 0.91 × (height [cm] - 152.4). The positive end-expiratory pressure (PEEP) was set at 10 cmH2O, with an inspiration-to-expiration ratio of 1:2, a respiratory rate of 16 breaths per minute, and an oxygen content of 41%
  Interventions: Device: VC Ventilation mode
- PRVC Ventilation mode group (Experimental): Group III patients received mechanical ventilation using the PRVC mode.The tidal volume during regulated breathing was determined based on the ideal body weight (IBW): 6-8 ml/kg (IBW for males: 50 + 0.91 × (height [cm] - 152.4); IBW for females: 45.5 + 0.91 × (height [cm] - 152.4). The positive end-expiratory pressure (PEEP) was set at 10 cmH2O, with an inspiration-to-expiration ratio of 1:2, a respiratory rate of 16 breaths per minute, and an oxygen content of 41%
  Interventions: Device: PRVC Ventilation mode

INTERVENTIONS:
Device: PC Ventilation mode — Patients were randomly assigned to three groups using a random number table and the random remainder grouping method at a ratio of 1:1:1. Group I received pressure control ventilation (PC).
  Arms: PC Ventilation mode group
Device: VC Ventilation mode — Patients were randomly assigned to three groups using a random number table and the random remainder grouping method at a ratio of 1:1:1. Group II received volume control ventilation (VC).
  Arms: VC Ventilation mode group
Device: PRVC Ventilation mode — Patients were randomly assigned to three groups using a random number table and the random remainder grouping method at a ratio of 1:1:1. Group III received pressure-regulated volume control ventilation (PRVC).
  Arms: PRVC Ventilation mode group

SUMMARY:
The goal of this clinical trial is to explore the clinical significance and value of the PRVC ventilation mode in Bariatric Surgery Patients. The main questions it aims to answer are：

* Do different ventilation patterns affect intracranial pressure and partial pressure of carbon dioxide in bariatric surgery patients?
* Does PRVC mode reduce intracranial pressure and partial pressure of carbon dioxide in bariatric surgery patients?
* Whether intracranial pressure can be quickly measured by monitoring a patient's optic nerve sheath diameter (ONSD)？ Researchers randomized bariatric surgery patients into PC, VC, and PRVC groups for comparison, looking at breathing mechanics, PaCO2, and ICP.

Participants will:

* take PC mode ventilation, VC mode ventilation, and PRVC mode ventilation
* monitor Respiratory mechanics, PaCO2, and ONSD

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective bariatric surgery.
* Age between 16 and 65 years.
* Continuous weight gain for more than 5 years with a BMI ≥ 35.
* ASA-PS (American Society of Anesthesiologists Physical Status) categorization of Grade II or III.

Exclusion Criteria:

* Patients who were dependent on alcohol or opioids.
* Patients with severe mental or intellectual disabilities.
* Patients with severe ocular conditions, such as ocular trauma, optic nerve tumors, or those wearing ocular prostheses.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
optic nerve sheath diameter [ONSD] | 1 year
  Patients were positioned supine with their eyes softly closed, and their eyes were protected with disposable transparent patches. A 7.5 MHz linear probe (Micromaxx Ultrasound System; SonoSite Inc., Bothell, WA, USA) was gently placed on the closed upper eyelid without applying pressure to the eyeball, and sufficient ultrasound gel was applied to ensure clear imaging. The optic nerve sheath was checked and measured 3 mm beyond the globe, and three ONSD measures were performed, with the average value utilized as the final ONSD measurement, which was accurate to 0.01 mm.
carbon dioxide partial pressure | 1 year
  Arterial blood carbon dioxide partial pressure, is an important indicator of alveolar ventilation, reflecting the respiratory factors in acid-base balance. Its reference value is usually 35-45 mmHg.
mean airway pressure (PAWM) | 1 year
  Mean airway pressure throughout the ventilation cycle
peak airway pressure (PAP) | 1 year
  Maximum pressure in the airway throughout inspiration
esophageal pressure (PES) | 1 year
  Esophageal manometry is the recording of pressure changes in various parts of the esophagus at rest and after swallowing, and is used to indicate the motor function of the upper and lower esophageal sphincters and the body of the esophagus, and to understand esophageal motility
tidal volume (TV) | 1 year
  Tidal volume is the volume of gas inhaled or exhaled each time when breathing calmly, it is an indicator to show lung volume, mainly used for ventilation function test in pulmonary function test. Tidal volume is the basis for assessing lung function and ventilation efficiency, and is an important indicator of lung volume
mean arterial pressure (MAP) | 1 year
  Mean arterial pressure is the average push given by the heart to blood flow throughout the cardiac cycle, with systolic pressure being the peak pressure and diastolic pressure being the pressure nadir.
heart rate (HR) | 1 year
  The normal adult heart rate ranges from 60 to 100 beats per minute, but infants and children have a faster heart rate than adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China